CLINICAL TRIAL: NCT04541420
Title: An Observational, Retrospective Study of Eribulin in Advanced Breast Cancer
Brief Title: Eribulin in mTNBC Patients
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Biyun Wang, MD, Professor, Fudan University
Other Study IDs: YOUNGBC-12
Record Dates: First submitted 2020-09-02; First posted 2020-09-09 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Breast Cancer
Keywords: Eribulin; TNBC
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Eribulin: Eribulin 1.4mg/m2 d1,8 iv q3w

SUMMARY:
To evaluate the efficacy and safety of Eribulin in patients with advanced breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced breast cancer included unresectable locally advanced breast cancer, de novo stage IV breast cancer, and recurrent metastatic breast cancer.
2. Eribulin treatment of advanced breast cancer for at least one cycle, between Dec 2019 and Aug 2020.
3. Available medical history.

Exclusion Criteria:

1. Incomplete medical history.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients diagnosed with breast cancer (according to International Classification of Diseases-10, ICD-10) with confirmed metastasis, regardless of being de novo diagnosed or progressed from a non-metastatic stage.
Sampling Method: Non-Probability Sample
Enrollment: 208 (Actual)
Dates: Start 2019-12-15 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2020-12-20 (Actual)

PRIMARY OUTCOMES:
PFS | 6 weeks
  Progression free survival
Adverse events | 6 weeks
  Number of participants with treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0)

CONTACTS AND LOCATIONS:
Overall Officials: Biyun Wang, Professor, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Shared information is not allowed by study cencer.